CLINICAL TRIAL: NCT04525755
Title: A Translational Randomized Clinical Trial of Varenicline Sampling to Promote Smoking Cessation and Scalable Treatment Dissemination
Brief Title: STARS (Smoking Treatment And Remote Sampling) Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Matthew Carpenter, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00098479
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Smoking; Smoking Cessation; Tobacco Smoking; Cigarette Smoking
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Smoking; Cigarette Smoking | interventions — Varenicline; Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1:1 ratio to receive a 4-week sample of varenicline, NRT, or not, with outcomes assessed through 12 weeks of follow-up. Participants in the varenicline sampling group will be given standard instructions on titration but ultimately will decide on their own as to if and how it is used. Dosing is lower than most industry trials of varenicline (1mg BID) but consistent with two trials of lower dosing that showed efficacy and with fewer side effects. Varenicline participants can choose to titrate 2mg if they wish, with shorter duration of sampling experience. Participants in NRT group will receive 28 day supply of nicotine patch (1patch x 28 days @ 14mg) and lozenge (14 per day x 28 days @4mg) with instructions to use based on number of cigarettes smoked per day. Like varenicline participants, smokers in NRT group can use as much or as little of the NRT as they wish.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Varenicline (.5mg BID) (Experimental): Participants will be randomized in a 2:1:1 ratio to receive a 4-week sample of varenicline (.5 mg, 60 tablets total), NRT, or not, with outcomes assessed through 12 weeks of follow-up. 324 participants will be enrolled in this group. Participants in the varenicline sampling group will be given standard instructions on titration but ultimately will decide on their own as to if and how it is used. Dosing is lower than most industry trials of varenicline (1mg BID) but consistent with two trials of lower dosing that showed efficacy and with fewer side effects. Varenicline participants can choose to titrate 2mg if they wish, with shorter duration of sampling experience.
  Interventions: Drug: Varenicline 0.5 MG
- Nicotine Replacement Therapy (NRT) (Active Comparator): Participants will be randomized in a 2:1:1 ratio to receive a 4-week sample of varenicline, NRT, or not, with outcomes assessed through 12 weeks of follow-up. 162 participants will be enrolled in this group. Participants in NRT group will receive 28 day supply of nicotine patch (1patch x 28 days @ 14mg) and lozenge (14 per day x 28 days @4mg) with instructions to use based on number of cigarettes smoked per day. Like varenicline participants, smokers in NRT group can use as much or as little of the NRT as they wish.
  Interventions: Drug: Nicotine Replacement Therapy (NRT)
- Control Group (No Intervention): Participants will be randomized in a 2:1:1 ratio to receive a 4-week sample of varenicline, NRT, or not, with outcomes assessed through 12 weeks of follow-up. 162 participants will be enrolled in this group.

INTERVENTIONS:
Drug: Varenicline 0.5 MG — varenicline comes in bottles of 56 - 0.5 mg pills
  Other Names: Chantix; Varenicline Pill
  Arms: Varenicline (.5mg BID)
Drug: Nicotine Replacement Therapy (NRT) — 28 day supply of nicotine patch (1 patch x 28 days @ 14 mg) and lozenge (14 per day x 28 days @ 4 mg)
  Other Names: NRT Sampling; Nicotine Patches and Lozenges; Nicotine Replacement Therapy Sampling; NRT
  Arms: Nicotine Replacement Therapy (NRT)

SUMMARY:
This is a research study to find out if a smoking cessation medications, either varenicline or nicotine replacement products (patches or lozenges), are effective when given to smokers, remotely, as a one-time sample.

Participants will either receive a sample of varenicline, nicotine patches and lozenges, or neither. This will be decided randomly. Participants have a 50%chance of receiving varenicline, a 25% chance of receiving nicotine products, and a 25% chance of receiving neither. If the participant is assigned to a group that receives free samples, they will be mailed to them free of charge. There is no requirement to use them, and it is completely up to the participants. There is also no requirement to quit in this study.

The study lasts for six months, and will involve six total surveys. In addition, investigators ask that participants complete daily diaries (about 1 minute each) for the first 4 weeks of the study. Both varenicline and nicotine replacement products are well-established medications that help smokers quit.

ELIGIBILITY:
Eligibility criteria include:

1. age 18+;
2. daily smoker (25+ days per previous month);
3. smoking 5+ cigarettes/day;
4. smoking > 1yr;
5. some interest in eventual quitting (>2 on 10-point scale);
6. has a primary care doctor and has seen that doctor at least once in past year;
7. not currently pregnant, breastfeeding, or planning to become pregnant;
8. no suicidal ideation in past month, nor any lifetime suicide attempt;
9. no reports of hallucinations;
10. no reports of history of seizures; nor cardiac/renal disease
11. own a smartphone or have regular (daily) access/use of email
12. if female, willing to take a pregnancy test
13. not currently taking any medications to help quit smoking
14. no diagnosis of schizophrenia or bipolar disorder
15. no members of the same household currently enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
7-day Quit Attempts | From study enrollment through end of six-month follow up
  Percentage of participants With 7-day self-reported point prevalence abstinence, among smokers randomized to a) varenicline, b) NRT, or c) no sampling control group

SECONDARY OUTCOMES:
Reduction in Smoking | At the week 4 follow up and week 26 follow up.
  Percentage of participants who have reduces their smoking by at least 50%, at both Week 4 and Week 26 follow-up, among smokers randomized to a) varenicline, b) NRT, or c) no sampling control group
Any Quit Attempts | From study enrollment through end of six-month follow up
  Any self-defined attempt to stop smoking cigarettes among smokers randomized to a) varenicline, b) NRT, or c) no sampling control group
Use of Smoking Cessation Medication | From study enrollment through end of six-month follow up
  Use of any smoking cessation medication among smokers randomized to a) varenicline, b) NRT, or c) no sampling control group

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT04525755/ICF_000.pdf